CLINICAL TRIAL: NCT02771418
Title: The Effects of Anaesthesia on Cerebral Oxygenation and Cognitive Function in Carotid Endarterectomy
Acronym: CEE-VIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Vsevolod V. Kuzkov, MD, PhD, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEE-VIMA
Record Dates: First submitted 2016-05-06; First posted 2016-05-13 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Endarterectomy; Postoperative Cognitive Dysfunction
Keywords: Carotid endarterectomy; postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIVA with propofol (Sham Comparator): Induction and maintenance of general anesthesia using TIVA with propofol
  Interventions: Drug: Propofol; Procedure: Elective carotid endarterectomy
- VIMA with sevoflurane (Active Comparator): Induction and maintenance of general anesthesia using VIMA with sevoflurane
  Interventions: Drug: Sevoflurane; Procedure: Elective carotid endarterectomy

INTERVENTIONS:
Drug: Propofol — Intravenous induction and maintenance of general anesthesia with propofol is a routine practice for this intervention
  Other Names: Tital intravenous anesthesia (TIVA)
  Arms: TIVA with propofol
Drug: Sevoflurane — Volatile induction and maintenance of general anesthesia with sevoflurane is a generally acceptable clinical approach for this intervention
  Other Names: Volatile induction and maintenance of anesthesia (VIMA)
  Arms: VIMA with sevoflurane
Procedure: Elective carotid endarterectomy

SUMMARY:
Volatile anesthetics interfere with cerebral blood flow and reperfusion-ischemia injury via the mechanism known as a preconditioning. A transient deterioration of local hemodynamics and oxygenation during carotid endarterectomy (CEE) might involve both hemispheres of brain and affect postoperative cognitive function. The goal of this study was to assess the effects of anesthetics on perioperative cerebral oxygenation and cognitive functions.

DETAILED DESCRIPTION:
Background: A transient deterioration of cerebral hemodynamics and oxygenation during CEE might involve both hemispheres of the brain and affects postoperative cognition. Despite some benefits of regional blocks, the majority of procedures of carotid endarterectomy (CEE) are performed under general anaesthesia. Surprisingly, the studies comparing the effects of sevoflurane and propofol on postoperative mental state in CEE are scarce and controversial. While propofol possesses some anti-inflammatory properties, volatile anesthetics can interfere with cerebral blood flow and reperfusion-ischaemia injury via the mechanism of pre- and postconditioning. The goal of this study is to assess the effects of the anesthetics on the perioperative cerebral oxygenation and cognitive functions in CEE.

Methods: The study and informed consent are approved by the Ethical Committee of the Northern State Medical University. Forty patients (males only) who are to undergo elective CEE will be included into a prospective study and randomised to two groups receiving either total intravenous anaesthesia (TIVA group, propofol + fentanyl) or the volatile induction and maintenance of anaesthesia (VIMA group, n = 20, sevoflurane + fentanyl). All patients were operated using temporary carotid bypass. Invasive arterial pressure (AP), gas exchange, and cerebral tissue oxygen saturation (SctO2, ForeSight, CAsMed, USA) over frontal region for ipsilateral (SctO2IPSI) and contralateral (SctO2CONTR) hemispheres were registered during the surgery and up to 20 hrs of the postoperative period. The cognitive changes will be assessed at 12 hrs before as well as on Days 1 and 5 after CEE by blinded investigator using Montreal Cognitive Assessment score (MoCA).

Data will be presented as median (25-75th percentiles). Intergroup comparison will be provided with Mann-Whitney U-test and correlation analysis with Spearman's coefficient (rho). P value below 0.05 was regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Male gender
* Informed consent
* Symptomatic carotid stenosis > 75%

Exclusion Criteria:

* Contralateral carotid occlusion
* Known allergy to the one of the compared medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Early postoperative cognitive dysfunction | 5 Days of the perioperative period
  Postoperative cognitive dysfunction assessed with MoCA score

SECONDARY OUTCOMES:
Cerebral desaturation | 0-20 hrs of the perioperative period
  Cerebral tissue oxygen saturation monitored intra- and postoperatively with non-invasive cerebral tissue oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- City hospital # 1 / Northern State Medical University,, Arkhangelsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Will be published in the peer-reviewed journal